CLINICAL TRIAL: NCT00693862
Title: Levodopa Concentration Profile After Repeated Doses of Stalevo
Brief Title: Pharmacokinetic Study With Repeated Doses of Stalevo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Jutta Hänninen, Clinical Study Manager, Orion Corporation, Orion Pharma
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2939115
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2008-06-09 (Estimated); Status verified 2008-06

CONDITIONS: Pharmacokinetics
Keywords: Focus of the study is pharmacokinetics of the study drug
MeSH Terms: interventions — Levodopa; Carbidopa; entacapone; carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stalevo (Experimental)
  Interventions: Drug: levodopa, carbidopa, entacapone
- levodopa/carbidopa (Active Comparator)
  Interventions: Drug: levodopa, carbidopa

INTERVENTIONS:
Drug: levodopa, carbidopa, entacapone
  Arms: Stalevo
Drug: levodopa, carbidopa
  Arms: levodopa/carbidopa

SUMMARY:
The purpose of this study is to show that higher minimum concentration values are obtained following repeated doses of Stalevo 4 times daily compared to lecodopa/carbidopa treatment with corresponding dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained
* Male or female patients with idiopathic Parkinson's disease with either a stable drug response or mild and predictable end-of-dose wearing-off symptoms.
* Hoehn and Yahr stage 1-2.5 performed during the "ON" state.
* Treatment with 3-5 daily doses of levodopa/DDCI ± entacapone with a total daily levodopa dose in the range of 300-600 mg.
* Unchanged levodopa/DDCI ± entacapone and other antiparkinsonian medication (dopamine agonists, monoamine oxidase B (MAO-B) inhibitor, amantadine and/or anticholinergics with doses recommended by the manufacturer), if any, for at least 2 weeks prior to the first treatment period.
* Age within 30-72 years, inclusive.

Exclusion Criteria:

* Secondary or atypical parkinsonism.
* Patients with moderate to marked wearing-off symptoms or any unpredictable "OFF"-periods.
* Patients with treatment-related peak-dose dyskinesia.
* Change in dose strength, daily dose or dosing frequency of any medicinal products used to treat other medical conditions than Parkinson's disease within 2 weeks.
* Use of any iron preparations or other chelating agents.
* Patients with a history of a laboratory abnormality consistent with, or clinically significant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, neurological or psychiatric disorder or any other major concurrent illness, which may influence the outcome of the study.
* History of neuroleptic malignant syndrome (NMS) and/or non-traumatic rhabdomyolysis, malignant melanoma, narrow-angle glaucoma or pheochromocytoma.
* Any abnormalities in laboratory values, vital signs or electrocardiogram (ECG) with clinical relevance.
* Patients using any antiparkinsonian drugs for rescue medication (including soluble levodopa formulations).
* Concomitant treatment with apomorphine, MAO-A inhibitors or non-selective MAO inhibitors.
* Known hypersensitivity to active substances or to any of the excipients of the study drugs.
* Participation in other drug studies within 60 days prior to study entry
* Unsuitable veins for repeated venopuncture.
* Blood donation or loss of significant amount of blood within 60 days prior to the screening.

Ages: 30 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-12; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | Blood samples collected frequently on day 4 of both periods

CONTACTS AND LOCATIONS:
Overall Officials: Jutta Hänninen, M.Sc., Study Director — Orion Corporation, Orion Pharma
Locations (3):
- Finland (3):
  - NEURO, Helsinki
  - Pharmacokinetics laboratory/Department of Pharmacology and Toxicology, Kuopio
  - Turku University Hospital, Turku